CLINICAL TRIAL: NCT01405014
Title: Pilot Study of the Hold Me Tight Relationship Enhancement Program With Couples Where One Partner Has an Acquired Brian Injury
Brief Title: Outcome Study of Hold Me Tight Program With Acquired Brian Injury (ABI) Populations
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NCTHMT-ABI
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2011-09

CONDITIONS: Marital Relationship
Keywords: Hold Me Tight; Emotionally Focused Therapy; Relationship enhancement; Couples counseling; Marital therapy; Acquired brain injury; Traumatic brain injury; Stroke
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Relationship enhancement group (Experimental): One group, all involved in the intervention
  Interventions: Behavioral: Hold Me Tight

INTERVENTIONS:
Behavioral: Hold Me Tight — Relationship enhancement group

SUMMARY:
The objectives of this research pilot project are to assess the efficacy of the Hold Me Tight Relationship Enhancement Program with couples where at least one partner has an acquired brain injury.

DETAILED DESCRIPTION:
Families, and spouses in particular, have been shown to play important roles in all aspects of health care, especially when family members are recovering from the trauma of sudden illness or an accident such as a brain injury. A limited body of evidence suggests couple therapy provides patients and their spouses with the opportunity to explore the experience of trauma as it relates to becoming physically disabled within the context of intimate relationships. Being in close contact and emotionally connected to a person who has experienced trauma becomes a chronic stressor that can cause family members to experience trauma symptoms themselves. This phenomenon is termed secondary traumatic stress. For example, children can mimic a parent's trauma responses through identification with the parent or direct training. This is a specific type of secondary traumatisation transmitted intergenerationally.

The research about individuals who have a traumatic brain injury (TBI) and the impact of the injury on family functioning has outlined a number of challenges including: psychological distress, particularly anxiety and depression, among caregivers; disruptions in family functioning; and the impact on relationships including caregiver burden. Furthermore, among the most difficult conditions for couples to deal with are those involving cognitive impairment.

Hold Me Tight is a couples enrichment program that is based on the Emotionally Focused Therapy (EFT) approach to working with couples. EFT is an empirically supported treatment that arose out of emotion theory and attachment theory. It views emotions as centrally important in the experience of self, in both adaptive and maladaptive functioning, and in therapeutic change. From the EFT perspective change occurs by means of awareness, regulation, reflection, and transformation of emotion taking place within the context of an empathetically attuned relationship. There is significant research on this approach and it has been found that 70-75% of couples move from distress to recovery and that the gains are sustained for months to years following the end of treatment. As such, EFT is an evidence based treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants must:
* be over the age of 18;
* be in a relationship at least 24 months and must be living together
* be at least 12 months post brain injury event
* be able to read and understand English, follow verbal instructions and provide verbal answers to questions;
* be able to follow-up as per Hold Me Tight program protocol;
* be willing to take part in the study, including completing all questionnaires before and after the intervention;
* are competent to give informed consent as determined by the Investigators

Exclusion Criteria:

* Participants must NOT:
* suffer from severe aphasia or dementia as determined by health chart;
* have active psychiatric illness;
* have other neurological condition(s);
* be couples where both partners have sustained a brain injury;
* have a high level of relationship distress better served by seeking individual couple therapy as indicated by a DAS score of 70 or less for either member of a couple

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Dyadic Adjustment Scale (DAS) | Change from Baseline in DAS scores at the end of the intervention and at three month follow-up
Beck Depression Inventory (BDI) | Change from Baseline in BDI scores at the end of the intervention and at three month follow-up
Beck Anxiety Inventory (BAI) | Change from Baseline in BAI scores at the end of the intervention and at three month follow-up

SECONDARY OUTCOMES:
Hold Me Tight Conversations Rating Scale | 12 weeks and three month follow-up
Hold Me Tight Program Evaluation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Allan, M.Ed., Principal Investigator — Dalhousie University
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada